CLINICAL TRIAL: NCT01333098
Title: Antiglucocorticoid Therapy for Cognitive Impairment in Late-life Anxiety Disorders
Acronym: Mifepristone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201011836
Record Dates: First submitted 2011-03-24; First posted 2011-04-11 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Anxiety Disorders
Keywords: anxiety; older adult; memory; cognitive; Saint Louis; treatment; cognitive impariment
MeSH Terms: conditions — Anxiety Disorders | interventions — Mifepristone

STUDY DESIGN:
Intervention Model Description: In the first week, participants were randomly assigned to mifepristone 300mg daily or placebo. In the subsequent 3 weeks, all participants received mifepristone 300mg.
Oversight: Data Monitoring Committee: No

ARMS (1):
- mifepristone (Experimental): 1 week mifepristone or placebo (followed by 3 weeks open label mifepristone)
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — 300mg per day, by mouth, for 21-28 days
  Other Names: Mifeprex; RU-486

SUMMARY:
This study seeks to develop and test a novel, mechanistic treatment for mitigating cognitive impairment in older adults with anxiety disorders. Anxiety disorders are common, severe, and disabling in older adults. One particularly impairing aspect of late-life anxiety disorders is cognitive impairment: impairments in memory and executive function cause disability, impede treatment response to psychotherapy, may lead to dementia, and are not corrected by standard anti-anxiety treatments.

This pilot study will test the glucocorticoid antagonist, mifepristone, for cognitive impairment in late-life anxiety disorders. Mifepristone blocks the effects of elevated cortisol levels on glucocorticoid receptors in the brain; it has been studied preliminarily in various neuropsychiatric disorders, such as psychotic depression and bipolar disorder, with well-documented safety and tolerability.

DETAILED DESCRIPTION:
Currently, no treatment exists to address cognitive impairment in late-life anxiety disorders. In this study, fifteen patients aged 60+ with an anxiety disorder (current or in partial remission) and subjective and/or objective evidence of cognitive impairment will receive treatment with mifepristone. At the baseline visit participants will be randomized to receive either mifepristone 300mg or a placebo daily for 7 days. Participants will be reassessed after 7 days (week 1 visit) of receiving study medication (mifepristone or placebo). At that time all participants will be provided mifepristone 300mg daily for the remaining 3 weeks of study treatment. The primary outcome measure will be neurocognition, as assessed by a battery of neuropsychological measures focusing on immediate and delayed memory and executive function (administered at baseline, week 1, week 4, and week 12). Saliva samples for cortisol measurement will be collected immediately following the baseline visit and week 4 visit. Secondary outcomes will be self-reported anxiety and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and older
* Non-demented by clinical evaluation
* Current or partially remitted generalized anxiety disorder or panic disorder
* Currently taking antidepressant treatment with stable dose for at least 8 weeks
* Memory impairment

Exclusion Criteria:

* Mild to severe dementia
* Diabetes
* Current alcohol or substance abuse
* Current or lifetime psychotic symptoms, bipolar disorder, or eating disorder
* Untreated endocrinologic disease
* Lifetime Cushing's or Addison's disease
* Current cancer
* History of metastatic cancer
* Current use of systemic corticosteroids

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Lenze, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lenze EJ, Hershey T, Newcomer JW, Karp JF, Blumberger D, Anger J, Dore P, Dixon D. Antiglucocorticoid therapy for older adults with anxiety and co-occurring cognitive dysfunction: results from a pilot study with mifepristone. Int J Geriatr Psychiatry. 2014 Sep;29(9):962-9. doi: 10.1002/gps.4085. Epub 2014 Mar 14. PMID 24633761

RESULTS

PARTICIPANT FLOW:
Groups:
- Mifepristone: 1 week mifepristone or placebo, followed by 3 weeks open label mifepristone
  Mifepristone: 300mg per day, by mouth, for 21-28 days
Period: Overall Study
Arm/Group | Mifepristone
Started | 15
Completed | 12
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Mifepristone: 1 week mifepristone or placebo followed by 3 weeks open label mifepristone
  Mifepristone: 300mg per day, by mouth, for 21-28 days
Arm/Group | Mifepristone
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Drug Acceptability, as Measured by Number of Participants With Dose-limiting Side Effects
Description: number of participants with dose-limiting side effects
Time Frame: Baseline, Week 2, Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone
Number analyzed (Participants) | 15
Participants | 1

2. Primary Outcome: Number of Participants With Self-reported Side Effects
Time Frame: 4 weeks
Measure: Number; unit: participants with reported side effects
Arm/Group | Mifepristone
Number analyzed (Participants) | 15
participants with reported side effects
  dizziness | 5
  fatigue | 3
  nausea | 2

3. Primary Outcome: Cognitive Changes Over Time, as Measured by Between Group and Within-subjects Comparison of Neuropsychological Measures.
Description: Memory composite z-score: The two memory measures were a 16-word list recall similar to the Rey auditory verbal learning test, which has been used by the Washington University Alzheimer's Disease Research Center; and two paragraphs from a set of paragraph recall tests validated as sensitive to effects of stress-level glucocorticoids. For each memory variable, a z score was computed for each participant, where z score = (participant score mean)/standard deviation. Then a single composite memory variable was created by summing up these z scores. Summed Z-scores range from -6 to 6, with scores above 0 being higher than the mean.
Time Frame: Baseline, Week 4, Week 12
Measure: Mean (Standard Error); unit: z-score
Groups:
- High Baseline Cortisol: baseline peak cortisol >6 ng/ml
- Without High Baseline Corisol: baseline peak cortisol <6 ng/ml
Arm/Group | High Baseline Cortisol | Without High Baseline Corisol
Number analyzed (Participants) | 5 | 8
z-score
  Baseline | 0.93 (1.58) | -0.59 (1.24)
  Week 4 | 1.85 (1.97) | -0.45 (1.34)
  Week 12 | 3.00 (2.20) | -0.26 (1.42)

4. Secondary Outcome: Anxiety Symptoms
Description: Self-report assessment of worry using Penn State Worry Questionnaire- Abbreviated, an 8-item measure (range 8-40 with high scores indicating higher levels of anxiety and worry symptoms.The average score for older adults with generalized anxiety disorder is 22, while the mean score for healthy older adults is 15.
Time Frame: baseline, week 4, week 12
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | High Baseline Cortisol | Without High Baseline Corisol
Number analyzed (Participants) | 5 | 8
Scores on a scale
  Baseline | 30.80 (4.27) | 27.88 (1.85)
  Week 4 | 22.40 (6.09) | 27.00 (1.51)
  Week 12 | 23.0 (6.02) | 25.29 (2.39)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the course of each participant's 12 week participation in the study which took place during a 4 month period.
Arm/Group | Mifepristone
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=15)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 2 (2)
Reduced T4 (Endocrine disorders) | 1 (1)
Worsening of pre-existing orthostatic hypotension (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes